CLINICAL TRIAL: NCT04178122
Title: Million Veteran Program Return of Actionable Results
Acronym: MVP-ROAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MVP030
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Results (Experimental): Participants in the Immediate Results arm will receive their genetic testing results from a genetic counselor at baseline following randomization.
  Interventions: Genetic: Result disclosure
- Delayed Results (Experimental): Participants in the Delayed Results arm will receive their genetic testing results from a genetic counselor 6 months after randomization.
  Interventions: Genetic: Result disclosure

INTERVENTIONS:
Genetic: Result disclosure — Disclosure of clinically confirmed, medically actionable genetic testing results and post-test genetic counseling session.

SUMMARY:
The purpose of the Million Veteran Program- Return of Actionable Results (MVP-ROAR) Study is to develop a process to return medically actionable genetic results to living MVP participants nationwide and to determine the impact of doing so on medical management and outcomes and Veteran quality of life.

DETAILED DESCRIPTION:
The Million Veteran Program - Return of Actionable Results (MVP-ROAR) Study is a randomized controlled trial of immediate vs. delayed (after 6 months) return of medically actionable, clinically confirmed genetic testing results. MVP participants with a medically actionable variant in their MVP chip genotype data will be contacted and offered the opportunity to receive clinical confirmation of this result through a research protocol. First, a non-randomized pilot trial will be conducted among 10 eligible MVP participants, followed by a randomized controlled trial of immediate vs. delayed clinical confirmation and reporting, delivered to participants nationwide via telegenetic counseling.

Three hypotheses will be tested:

Hypothesis 1 (LDL-C change): LDL-C reduction after 6 months will be greater in the Immediate Results arm compared to the Delayed Results arm (primary outcome) Hypothesis 2 (LDL-C target): The proportion of participants meeting clinically significant LDL-C targets (<100mg/dL for primary prevention and <70 mg/dL for secondary prevention) at 6 months will be greater in the Immediate Results arm than in the Delayed Results arm (secondary outcome) Hypothesis 3 (Pharmacotherapy): the proportion of participants with an intensification of lipid-lowering pharmacotherapy will be greater in the Immediate Results arm than in the Delayed Results arm (secondary outcome)

ELIGIBILITY:
Inclusion Criteria:

* Living enrollee in MVP
* Is identified to have a pathogenic or likely pathogenic variant in the gene(s) of interest in MVP genotype data

Exclusion Criteria:

* Previously underwent genetic testing for the condition of interest
* Is incarcerated
* Is pregnant

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Vassy, MD MPH, Study Chair — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual-level trial data through a data repository housed on a secure VA server and accessible only to outside investigators with IRB and other regulatory approvals. MVP ROAR Study data will also be stored in the VA MVP Central Database.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Vassy JL, Brunette CA, Yi T, Assimes TL, Christensen KD, Knowles JW, Sturm AC, Sun YV, Alexander N, Cardellino MP, Harrison A, Gerety HL, Pyatt M, Vered R, Wilson PWF, Natarajan P, Whitbourne SB, Gaziano JM, Muralidhar S, Danowski ME; Veterans Affairs Million Veteran Program. Opportunistic Genomic Screening for Familial Hypercholesterolemia to Improve Low-Density Lipoprotein Cholesterol: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2549664. doi: 10.1001/jamanetworkopen.2025.49664. PMID 41511773
- [Derived] Vassy JL, Brunette CA, Yi T, Harrison A, Cardellino MP, Assimes TL, Christensen KD, Devineni P, Gaziano JM, Gong X, Hui Q, Knowles JW, Muralidhar S, Natarajan P, Pyarajan S, Sears MG, Shi Y, Sturm AC, Whitbourne SB, Sun YV, Danowski ME; Million Veteran Program. Design and pilot results from the Million Veteran Program Return Of Actionable Results (MVP-ROAR) Study. Am Heart J. 2024 Oct;276:99-109. doi: 10.1016/j.ahj.2024.04.021. Epub 2024 May 17. PMID 38762090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on February 27, 2020. 459 MVP participants with a suspected FH-associated variant were recruited and assessed for eligibility.
Pre-assignment Details: 347 participants were excluded from randomization due to: not meeting inclusion criteria, unable to contact, declined to participate, lost to follow up, withdrew, or deceased.
Period: Overall Study
Arm/Group | Immediate Results | Delayed Results
Started | 55 | 57
Completed | 49 | 43
Not Completed | 6 | 14
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 2 | 0
Not completed — Did not complete testing | 3 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Results | Delayed Results | Total
Number analyzed (Participants) | 55 | 57 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (14.1) | 65.2 (12.6) | 65.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 44 | 50 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 19 | 31
  White | 39 | 33 | 72
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 51 | 50 | 101
  Unknown or Not Reported | 0 | 1 | 1
LDL-C [Mean (Full Range); unit: mg/dL] | 114.4 [22 to 376] | 104.7 [2 to 274] | 109.5 [2 to 376]

OUTCOME MEASURES:

1. Primary Outcome: LDL-C Change
Description: Change in LDL-C after 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Results | Delayed Results
Number analyzed (Participants) | 55 | 57
mg/dL | -8.0 (32.3) | 2.4 (28.9)

2. Secondary Outcome: LDL-C Target
Description: The number of participants meeting clinically significant LDL-C targets (< 100mg/dL for primary prevention and <70 mg/dL for secondary prevention) at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Results | Delayed Results
Number analyzed (Participants) | 55 | 57
Participants | 15 | 14

3. Secondary Outcome: Pharmacotherapy
Description: The number of participants with an intensification of lipid-lowering pharmacotherapy, a composite outcome including prescription of new monotherapy, dose escalation of existing pharmacotherapy, and addition of one or more medications to existing pharmacotherapy.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Results | Delayed Results
Number analyzed (Participants) | 55 | 57
Participants | 11 | 5

4. Other Pre Specified Outcome: Cascade Testing
Description: The number of first-degree relatives having undergone genetic testing at 6 months.
Time Frame: 6 months
Population: Only the participants in the immediate results arm completed this survey measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Results | Delayed Results
Number analyzed (Participants) | 55 | 0
Participants | 3 | 0

5. Other Pre Specified Outcome: Lifestyle Behaviors
Description: The number of participants reporting healthy lifestyle behaviors (smoking, physical activity, and saturated fat intake) at 6 months, measured by questionnaire responses.
Time Frame: 6 months
Population: Survey responses fully or partially missing from some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Results | Delayed Results
Number analyzed (Participants) | 55 | 57
Participants
  6-month physical activity: number analyzed (Participants) | 50 | 44
  6-month physical activity: YES, I have been for MORE than 6 months | 30 | 27
  6-month physical activity: YES, I have, but for less than 6 months | 3 | 4
  6-month physical activity: NO, but I intend to in the next 30 days | 4 | 6
  6-month physical activity: NO, but I intend to in the next 6 months | 6 | 1
  6-month physical activity: NO, and I do NOT intend to in the next 6 months | 7 | 6
  6-month saturated fat consumption: number analyzed (Participants) | 48 | 44
  6-month saturated fat consumption: YES, I have been for MORE than 6 months | 23 | 28
  6-month saturated fat consumption: YES, I have, but for less than 6 months | 2 | 0
  6-month saturated fat consumption: NO, but I intend to in the next 30 days | 1 | 3
  6-month saturated fat consumption: NO, but I intend to in the next 6 months | 3 | 0
  6-month saturated fat consumption: NO, and I do NOT intend to in the next 6 months | 19 | 13

6. Other Pre Specified Outcome: Quality of Life (Veterans RAND Survey)
Description: Quality of life, measured by the Veterans RAND (distributed by RAND Corporation) 12-item Health Survey (VR-12). Items are scored using an algorithm and summarized into two scores (Physical Component Score and a Mental Component Score) ranging from 0-100, with a higher score indicating better health.
Time Frame: 6 months
Population: Survey responses fully or partially missing from some participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Results | Delayed Results
Number analyzed (Participants) | 55 | 54
score on a scale
  Physical component: baseline | 38.32 (11.05) | 39.08 (14.47)
  Physical component: 6-month: number analyzed (Participants) | 49 | 44
  Physical component: 6-month | 39.10 (11.44) | 40.58 (14.14)
  Physical component: change: number analyzed (Participants) | 49 | 44
  Physical component: change | 0.78 (4.45) | 1.5 (4.83)
  Mental component: baseline | 47.78 (13.98) | 49.69 (12.98)
  Mental component: 6-month: number analyzed (Participants) | 49 | 44
  Mental component: 6-month | 47.38 (14.29) | 49.99 (12.98)
  Mental component: change: number analyzed (Participants) | 49 | 44
  Mental component: change | -0.403 (6.29) | 0.31 (4.66)

7. Other Pre Specified Outcome: Medication Adherence
Description: Medication adherence at 6 months, measured by the Beliefs About Medicines Questionnaire (BMQ).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Results | Delayed Results
Number analyzed (Participants) | 55 | 57
Participants
  Doctors use too many medications: Strongly agree | 8 | 6
  Doctors use too many medications: Agree | 24 | 14
  Doctors use too many medications: Disagree | 12 | 18
  Doctors use too many medications: Strongly disagree | 1 | 0
  Doctors use too many medications: Neither agree nor disagree | 5 | 7
  Doctors use too many medications: Did not respond/ Missing | 5 | 12
  People who take medicines should stop their treatment every now and then: Strongly agree | 0 | 0
  People who take medicines should stop their treatment every now and then: Agree | 3 | 0
  People who take medicines should stop their treatment every now and then: Disagree | 30 | 32
  People who take medicines should stop their treatment every now and then: Strongly disagree | 16 | 10
  People who take medicines should stop their treatment every now and then: Neither agree nor disagree | 1 | 3
  People who take medicines should stop their treatment every now and then: Did not respond/ Missing | 5 | 12
  If doctors have more time with patients they would prescribe fewer medicines: Strongly agree | 6 | 2
  If doctors have more time with patients they would prescribe fewer medicines: Agree | 20 | 18
  If doctors have more time with patients they would prescribe fewer medicines: Disagree | 10 | 15
  If doctors have more time with patients they would prescribe fewer medicines: Strongly disagree | 3 | 1
  If doctors have more time with patients they would prescribe fewer medicines: Neither agree nor disagree | 11 | 9
  If doctors have more time with patients they would prescribe fewer medicines: Did not respond/ Missing | 5 | 12
  Doctors place too much trust in medicines: Strongly agree | 7 | 3
  Doctors place too much trust in medicines: Agree | 22 | 17
  Doctors place too much trust in medicines: Disagree | 12 | 15
  Doctors place too much trust in medicines: Strongly disagree | 3 | 0
  Doctors place too much trust in medicines: Neither agree nor disagree | 6 | 10
  Doctors place too much trust in medicines: Did not respond/ Missing | 5 | 12
  Medicines do more harm than good: Strongly agree | 2 | 1
  Medicines do more harm than good: Agree | 6 | 3
  Medicines do more harm than good: Disagree | 24 | 25
  Medicines do more harm than good: Strongly disagree | 10 | 9
  Medicines do more harm than good: Neither agree nor disagree | 8 | 7
  Medicines do more harm than good: Did not respond/ Missing | 5 | 12
  Most medicines are addictive: Strongly agree | 1 | 1
  Most medicines are addictive: Agree | 6 | 5
  Most medicines are addictive: Disagree | 33 | 32
  Most medicines are addictive: Strongly disagree | 6 | 6
  Most medicines are addictive: Neither agree nor disagree | 4 | 1
  Most medicines are addictive: Did not respond/ Missing | 5 | 12
  All medicines are poisons: Strongly agree | 1 | 0
  All medicines are poisons: Agree | 0 | 0
  All medicines are poisons: Disagree | 34 | 28
  All medicines are poisons: Strongly disagree | 14 | 16
  All medicines are poisons: Neither agree nor disagree | 1 | 1
  All medicines are poisons: Did not respond/ Missing | 5 | 12
  Natural remedies are safer than medicines: Strongly agree | 2 | 2
  Natural remedies are safer than medicines: Agree | 11 | 5
  Natural remedies are safer than medicines: Disagree | 14 | 20
  Natural remedies are safer than medicines: Strongly disagree | 7 | 3
  Natural remedies are safer than medicines: Neither agree nor disagree | 16 | 15
  Natural remedies are safer than medicines: Did not respond/ Missing | 5 | 12

8. Other Pre Specified Outcome: Smoking Status
Description: 6-month smoking status
Time Frame: 6-month
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Results | Delayed Results
Number analyzed (Participants) | 50 | 44
Participants
  Never smoked | 15 | 23
  Quit > 6 months | 30 | 16
  Quit within 6 months | 1 | 2
  Current smoker | 4 | 3

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not systematically assessed for the study.
Arm/Group | Immediate Results | Delayed Results
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limitations include:

1. Lower enrollment than planned
2. Baseline LDL-C values were carried forward for 15 participants missing their 6-month value
3. Participants with variants only detectable by sequencing were not included
4. LDL-C is a surrogate endpoint for long-term clinical outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT04178122/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT04178122/SAP_001.pdf